CLINICAL TRIAL: NCT01779791
Title: An Open-Label, Multicenter, Single-Arm, Phase 2 Study of PCI-32765 (Ibrutinib) in Subjects With Refractory Follicular Lymphoma
Brief Title: A Study of PCI-32765 (Ibrutinib) in Patients With Refractory Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100956; 2012-004097-26 (EudraCT Number); PCI-32765FLR2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-01-25; First posted 2013-01-30 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Lymphoma
Keywords: Lymphoma; Refractory follicular lymphoma; Chemoimmunotherapy-resistant follicular lymphoma; PCI-32765; Ibrutinib; IMBRUVICA
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PCI-32765 (Ibrutinib) (Experimental)
  Interventions: Drug: PCI-32765 (Ibrutinib)

INTERVENTIONS:
Drug: PCI-32765 (Ibrutinib) — 560 mg capsules administered orally once daily, continuously on a 21-day cycle until progressive disease.
  Other Names: IMBRUVICA

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PCI-32765 (ibrutinib) administered to patients with chemoimmunotherapy-resistant follicular lymphoma (FL).

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) study of PCI-32765 (ibrutinib) in approximately 110 patients with chemoimmunotherapy-resistant FL whose disease has relapsed from at least 2 prior lines of therapy, including at least 1 rituximab combination chemotherapy regimen. Each patient must have resistant disease to the last therapy (defined as progression of disease [PD] during or within 12 months of the last dose of chemotherapy in a CD20 antibody combination chemotherapy regimen). The study will include the following phases: screening (up to 30 days prior to the first dose of study drug), treatment (until PD or unacceptable toxicity), and posttreatment follow-up (until death, lost to follow up, withdrawal of consent, or study end [defined as 2 years after the last patient is enrolled]). Patients will receive 560 mg of PCI-32765 by mouth once daily on a 21-day cycle. Treatment will be continuous (without interruption) and self-administered at home. The treatment phase will extend from administration of the first dose of study medication until PD or unacceptable toxicity. If a patient who had radiological evidence of PD is clinically stable or improving or exhibiting signs of tumor flare without confirmation of PD by PET or biopsy, they may continue treatment with ibrutinib upon request by the investigator and approval by the sponsor. Posttreatment follow-up will extend from the end of treatment until death, lost to follow up, withdrawal of consent, or study end. Every patient, except for those who explicitly withdraw consent from further site contact, will be followed for survival status until the study ends. In addition, data on subsequent antineoplastic therapy will also be collected. Serial pharmacokinetic samples will be collected and efficacy and safety will be monitored throughout the study. A separate assessment of pharmacokinetics is planned for patients who receive a strong or moderate CYP3A4/5 inhibitor while receiving treatment with ibrutinib. For patients who have already discontinued ibrutinib due to PD, have taken no other anticancer therapy, and now have a radiologically documented delayed response, resumption of ibrutinib is permitted on a case-by-case basis, upon request by the investigator and approval of the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of Grade 1, 2, or 3a follicular lymphoma (FL) without clinical or pathological evidence of transformation
* Previously treated with at least 2 prior lines of therapy, including at least 1 rituximab combination chemotherapy regimen; last prior line of therapy includes an anti CD20 monoclonal antibody-containing chemotherapy regimen (separate lines of therapy are defined as different regimens that are either separated by disease progression, refractory disease, or relapsed disease)
* Resistant disease to the last therapy, defined as progression of disease during or within 12 months of the last dose of chemotherapy in a CD20 antibody combination chemotherapy regimen
* At least 1 measurable site of disease according to International Working Group Revised Response Criteria for Malignant Lymphoma
* Eastern Cooperative Oncology Group performance status grade 0 or 1
* Hematology and biochemical laboratory values must be within protocol-defined parameters within 7 days prior to enrollment
* Agrees to protocol-defined use of effective contraception
* Women of childbearing potential must have a negative serum or urine pregnancy test at screening

Exclusion Criteria:

* Prior nitrosoureas within 6 weeks, chemotherapy within 3 weeks, therapeutic anticancer antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy or other investigational agents within 3 weeks, or major surgery within 4 weeks of first dose of study drug
* Prior treatment with PCI-32765 or other Bruton's tyrosine kinase inhibitors (patients who progressed or became refractory while on treatment with PI3K inhibitors are excluded)
* Concurrent enrollment in another therapeutic investigational clinical treatment study
* Received a prior allogeneic hematopoietic stem cell transplant (prior autologous hematopoietic stem cell transplant is allowed)
* Known central nervous system lymphoma
* History of prior malignancy (except malignancy treated with curative intent and with no known active disease present for >=3 years before enrollment, adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, or adequately treated cervical carcinoma in situ without evidence of disease)
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong cytochrome P450 (CYP)3A4/5 inhibitors
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Known history of Human Immunodeficiency Virus (HIV) or active infection with Hepatitis C or active infection with Hepatitis B or any uncontrolled active systemic infection requiring intravenous antibiotics
* Women who are pregnant or breastfeeding
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of PCI-32765 capsules, or put the study outcomes at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-04-17 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2016-05-18 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 2 years after the last patient is enrolled

SECONDARY OUTCOMES:
Duration of response | Every 12 weeks during the first 96 weeks, followed by every 24 weeks thereafter until disease progression (up to 2 years after the last patient is enrolled)
Progression-free survival | Up to progressive disease, death, lost to follow-up, withdrawal of consent, or study end (up to 2 years after the last patient is enrolled)
Overall survival | Up to death, lost to follow-up, withdrawal of consent, or study end (up to 2 years after the last patient is enrolled)
Time to response | Every 12 weeks during the first 96 weeks, followed by every 24 weeks thereafter until disease progression (up to 2 years after the last patient is enrolled)
Number of patients experiencing resolution of lymphoma-related B symptoms | Day 1 of every cycle during the first 12 months, thereafter every other cycle (up to 2 years after the last patient is enrolled)
Number of patients identified with blood biomarkers that alter B-cell receptor signaling or activate alternative signaling pathways | Day 1 of Cycles 1-3, and time of disease progression, or at end-of treatment visit for patients who discontinue treatment without disease progression
Minimum plasma concentration of PCI-32765 | Pre-dose Day 1 of Cycles 1-3, post-dose Day 1 of Cycles 1, 2 at 1, 2, and 4 hours
Oral plasma clearance of PCI-32765 | Pre-dose Day 1 of Cycles 1-3, post-dose Day 1 of Cycles 1, 2 at 1, 2, and 4 hours
Oral volume of distribution at steady state of PCI-32765 | Pre-dose Day 1 of Cycles 1-3, post-dose Day 1 of Cycles 1, 2 at 1, 2, and 4 hours
Area under the plasma-concentration time curve of PCI-32765 | Pre-dose Day 1 of Cycles 1-3, post-dose Day 1 of Cycles 1, 2 at 1, 2, and 4 hours
Number of participants affected by an adverse event | Up to 30 days after the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (54):
- United States (20):
  - Los Angeles, California
  - Stanford, California
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Chicago, Illinois
  - Westwood, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Detroit, Michigan
  - Hackensack, New Jersey
  - New Brunswick, New Jersey
  - New York, New York
  - Greenville, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - Burlington, Vermont
  - Seattle, Washington
- Australia (5):
  - Adelaide
  - Concord
  - Melbourne
  - Milton
  - Prahran
- Belgium (3):
  - Courrière
  - Ghent
  - Leuven
- France (7):
  - Créteil
  - Nice
  - Nîmes
  - Paris
  - Pessac
  - Pierre-Bénite
  - Rennes
- Germany (4):
  - Cologne
  - Heidelberg
  - Mainz
  - Ulm
- Poland (3):
  - Krakow
  - Warsaw
  - Wroclaw
- Russia (5):
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Volgograd
  - Yekaterinburg
- Spain (3):
  - Barcelona
  - Marbella
  - Salamanca
- United Kingdom (4):
  - Liverpool
  - London
  - Manchester
  - Southampton

REFERENCES:
- [Derived] Balasubramanian S, Hodkinson B, Schuster SJ, Fowler NH, Trotman J, Hess G, Cheson BD, Schaffer M, Sun S, Deshpande S, Vermeulen J, Salles G, Gopal AK. Identification of a genetic signature enriching for response to ibrutinib in relapsed/refractory follicular lymphoma in the DAWN phase 2 trial. Cancer Med. 2022 Jan;11(1):61-73. doi: 10.1002/cam4.4422. Epub 2021 Nov 17. PMID 34791836
- [Derived] Gopal AK, Schuster SJ, Fowler NH, Trotman J, Hess G, Hou JZ, Yacoub A, Lill M, Martin P, Vitolo U, Spencer A, Radford J, Jurczak W, Morton J, Caballero D, Deshpande S, Gartenberg GJ, Wang SS, Damle RN, Schaffer M, Balasubramanian S, Vermeulen J, Cheson BD, Salles G. Ibrutinib as Treatment for Patients With Relapsed/Refractory Follicular Lymphoma: Results From the Open-Label, Multicenter, Phase II DAWN Study. J Clin Oncol. 2018 Aug 10;36(23):2405-2412. doi: 10.1200/JCO.2017.76.8853. Epub 2018 May 31. PMID 29851546
- See also: An Open-label, Multicenter, Single-arm, Phase 2 Study of PCI-32765 (ibrutinib) in Subjects with Refractory Follicular Lymphoma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3624&filename=CR100956_CSR.pdf